CLINICAL TRIAL: NCT00118378
Title: Modafinil Treatment for Fatigue in HIV+ Patients
Brief Title: Effectiveness of Modafinil for Treating Fatigue in Adults With HIV/AIDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #4839; R01MH072383-01 (NIH); DAHBR 9A-ASNM
Record Dates: First submitted 2005-07-06; First posted 2005-07-11 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections; Fatigue
Keywords: HIV; AIDS; Modafinil; Depression
MeSH Terms: conditions — HIV Infections; Fatigue; Acquired Immunodeficiency Syndrome; Depression | interventions — Modafinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modafinil (Experimental): Participants will take modafinil for 4 weeks.
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Participants will take placebo for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — 50 mg per day, increasing to 200 mg per day as clinically indicated
  Other Names: Provigil
  Arms: Modafinil
Drug: Placebo — 50 mg per day, increasing to 200 mg per day as clinically indicated
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This study will determine whether modafinil (Provigil®), a medication approved for the treatment of narcolepsy, is effective in reducing fatigue in adults with HIV/AIDS.

DETAILED DESCRIPTION:
Fatigue is a common problem for many people with HIV/AIDS, interfering with daily activities and serving as a significant barrier to working among those whose health is otherwise stable or restored by antiretroviral (ARV) medication. Fatigue in HIV is associated with disability and diminished quality of life. It may be caused by ARVs or by the virus itself. This study will determine if modafinil can reduce fatigue in HIV/AIDS patients.

This study will last 12 weeks. Participants will be randomly assigned to receive either modafinil or placebo daily for 4 weeks. Participants who show an improvement in symptoms will receive modafinil for an additional 8 weeks. Participants who do not respond to modafinil will have the opportunity to receive other drug treatments. All participants will have weekly study visits for the first 4 weeks of the study and biweekly visits for the remainder of the study. At each visit, participants will complete various tasks to determine cognitive function and self-report scales will be used to determine symptoms of depression and fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75
2. HIV+
3. Clinically significant fatigue (score of 4.5+ on Fatigue Severity Scale, plus impairment on 1+ categories of Role Function Scale)
4. Fatigue duration for 3+ months
5. English-speaking
6. Able to give informed consent
7. Fecund women uses barrier method of contraception

Exclusion Criteria:

1. Primary care doctor does not approve of study participation
2. Unstable medical condition (e.g. liver failure;cirrhosis, new onset opportunistic infection [O.I.] in past month)
3. Untreated hypogonadism, except for men for whom testosterone replacement is medically contraindicated (serum testosterone below the reference range)
4. Untreated hypothyroidism (thyroid stimulating hormone [TSH] over 5 IUI/mL)
5. Untreated and uncontrolled hypertension
6. Clinically significant anemia (hematocrit <30%)
7. Started testosterone or nandrolone in past 6 weeks
8. Started or changed an antiretroviral regimen in past 4 weeks if fatigue predated the change; otherwise, started or changed regimen in past 2 months
9. Untreated or under-treated major depressive disorder
10. Started antidepressant medication within past 6 weeks
11. Substance abuse/dependence (past 4 months)
12. Regular and frequent cannabis use (> twice/week regularly)
13. Currently clinically significant suicidal ideation or Hamilton Depression Rating Scale (HAM-D) >24
14. History or current psychosis or bipolar disorder
15. Pregnant or breastfeeding
16. Significant untreated insomnia (score >3 on HAM-D insomnia items)
17. Currently taking psychostimulant medication or past nonresponse to modafinil
18. Has no alternative viable antiretroviral regimen after the current one
19. Left ventricular hypertrophy; mitral valve prolapse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2004-12; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G. Rabkin, PhD, MPH, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Rabkin JG, McElhiney MC, Rabkin R, Ferrando SJ. Modafinil treatment for fatigue in HIV+ patients: a pilot study. J Clin Psychiatry. 2004 Dec;65(12):1688-95. doi: 10.4088/jcp.v65n1215. PMID 15641875
- [Result] Rabkin JG, McElhiney MC, Rabkin R, McGrath PJ. Modafinil treatment for fatigue in HIV/AIDS: a randomized placebo-controlled study. J Clin Psychiatry. 2010 Jun;71(6):707-15. doi: 10.4088/JCP.09m05171bro. Epub 2010 May 4. PMID 20492840
- See also: Click here for a related study currently recruiting participants. — http://clinicaltrials.gov/ct2/show/NCT00737204?term=rabkin&rank=4

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from January 2005 until December 2008.
Groups:
- Modafinil: Participants will take modafinil for 4 weeks. If responsive, participants will be offered 8 additional weeks of modafinil.
- Placebo: Participants will take placebo for 4 weeks, if not responsive, a 12-week course of modafinil will be offered.
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 62 | 53
Completed | 60 | 45
Not Completed | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 62 | 53 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 53 | 113
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.94 (9.35) | 45.74 (8.57) | 45.84 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 54 | 46 | 100
Region of Enrollment [Number; unit: participants]
  United States | 62 | 53 | 115

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Severity Scale (FSS)
Description: The FSS is a 9-item self-report scale that measures the impact of fatigue on everyday functioning. Each item is rated on a scale of 1 to 7. Total scores range from 9 to 63, with a higher value indicating greater impairment due to fatigue.
Time Frame: Measured at baseline and Week 4
Population: The WEEK 4 outcome analyses are based on an intention to treat sample which includes the 10 dropouts (2 on Modafinil and 8 on Placebo), using the last data point brought forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Modafinil: Participants randomized to modafinil for 4 weeks. If responsive, participants will be offered 8 additional weeks of modafinil.
- Placebo: Participants randomized to placebo for 4 weeks, if not responsive, a 12-week course of modafinil will be offered.
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 62 | 53
units on a scale
  Baseline FSS | 52 (7) | 52 (6)
  Week 4 FSS | 34 (5) | 43 (13)
Statistical Analysis 1: Comparison: Modafinil vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Primary Outcome: Role Function Scale Outcome
Description: The Role Function Scale includes 10 items drawn from the Short Form 36-item Health Survey (SF-36) and other SF versions. It is intended to assess the extent to which fatigue has a behavioral impact on daily activities. Scores of frequency in the past week, on a 5-point scale, are summed with higher scores signifying greater role impairment. Scores range from 10 to 50.
Time Frame: Measured at baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 62 | 53
units on a scale
  Baseline Role Function Scale | 39 (7) | 36 (6)
  Week 4 Role Function Scale | 22 (9) | 27 (11)
Statistical Analysis 1: Comparison: Modafinil vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Secondary Outcome: CD4 Cell Count
Description: CD4 cell count is a laboratory marker providing an indication of immune functioning. Blood was drawn for this measure at baseline and week 4. The reference range for CD4 cell count is 490-1740, and a clinically significant change is defined as a change of >= 100 cells. A higher number is associated with better immune functioning.
Time Frame: Measured at baseline and Week 4
Population: Results were included for patients on whom baseline and week 4 labs were drawn.
Measure: Mean (Standard Deviation); unit: Cells/mcL
Groups:
- Modafinil: Participants randomized to modafinil for 4 weeks.
- Placebo: Participants randomized to placebo for 4 weeks.
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 58 | 44
Cells/mcL
  Baseline CD4 cell count | 481 (249) | 459 (257)
  Week 4 CD4 cell count | 466 (244) | 482 (240)
Statistical Analysis 1: Comparison: Modafinil vs Placebo; Week 4 CD4 cell count; Test type: Superiority or Other; p = .150, ANOVA

4. Secondary Outcome: HIV RNA Viral Load
Description: HIV RNA viral load assay is a laboratory measure indicating viral activity. Because of the large range of possible values (50-100,000 copies), this measure is presented in log10. We entered the log10 value of 1.69 when the laboratory result stated "under 50 copies," which was the assay's lowest limit of detectability during the study.
Time Frame: Measured at baseline and Week 4
Population: Results were included for patients on whom baseline and week 4 labs were drawn.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 58 | 44
Log10 copies/mL
  Baseline Log10 Viral Load | 2.53 (1.2) | 2.41 (1.2)
  Week 4 Log10 Viral load | 2.31 (1.0) | 2.30 (1.1)
Statistical Analysis 1: Comparison: Modafinil vs Placebo; Test type: Superiority or Other; p = .459, ANOVA

ADVERSE EVENTS:
Time Frame: Weeks 1-4 during the double-blind phase of the study.
Arm/Group | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/53
Other Adverse Events (participants affected / at risk) | 0/62 | 0/53

LIMITATIONS AND CAVEATS:
This study was conducted at a single site in an urban setting where most patients have good access to medical care. Women were under-represented despite outreach efforts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes